CLINICAL TRIAL: NCT03662906
Title: The Efficacy and Safety of Electroacupuncture for Urinary Function of Patients With CUR Secondary to Lower Motor Neuron Lesion: A Multi-center Randomized Sham-controlled Trial
Brief Title: Electroacupuncture for Patients With Chronic Urinary Retention Secondary to Lower Motor Neuron Lesion
Acronym: CUR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liu Zhishun, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-102-KY-01
Record Dates: First submitted 2018-09-06; First posted 2018-09-10 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Chronic Urinary Retention
Keywords: Chronic urinary retention; Electroacupuncture; Urinary function; Randomized controlled trial
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture (Experimental): Bilateral Shenshu (BL23), Ciliao (BL32), Zhongliao (BL33), Huiyang (BL35), and Sanyinjiao (SP6) will be inserted by the needles (0.30 mm in diameter, 75 mm in length or 0.40 mm diameter, 100 mm in length, Hwato Brand, Suzhou Medical Appliance Factory, China).
  Interventions: Other: Electroacupuncture
- Sham electroacupuncture (Sham Comparator): Sham Bilateral Shenshu (BL23), Ciliao (BL32), Zhongliao (BL33), Huiyang (BL35), and Sanyinjiao (SP6) will be inserted by the needles (0.20 mm in diameter, 25 mm in length, Hwato Brand, Suzhou Medical Appliance Factory, China).
  Interventions: Other: Sham electroacupuncture

INTERVENTIONS:
Other: Electroacupuncture — Bilateral BL32 and BL 33 will be inserted to a depth of 70-95 mm with an angle of 20-30° inward and downward into the second and third sacral foramen. Bilateral BL35 will be inserted to a depth of 60-70 mm with a slightly superolateral direction using needles (0.30 mm in diameter, 75 mm in length). Bilateral BL23 and SP6 will be inserted vertically to a depth of 25-30 mm using needles (0.30 mm in diameter, 40 mm in length). The electric stimulators (6805-D electroacupuncture apparatus, Guangzhou Jiayu Medical Company, China) will connect the bilateral BL32, BL33, BL35 and SP 6 and a continuous wave of 10 Hz frequency and an intensity of 5-10 mA for BL 32 and BL 33 and an intensity of 1-5 mA for SP 6 will be applied.
  The needles will be retained for 60 mins for each treatment session. The participants will be treated three times a week, on alternate days, for 12 successive weeks; 18 sessions for each patient in total.
  Arms: Electroacupuncture
Other: Sham electroacupuncture — Sham BL 23, BL32 and BL33 which are 2 cm lateral to BL23, BL33 and BL35 will be inserted by the needles (0.20 mm in diameter, 25 mm in length) to a depth of 2-3 mm. Sham SP 6 which is at the midpoint between the spleen meridian and the kidney meridian will be inserted by the needles (0.20 mm in diameter, 25 mm in length) to a depth of 2-3 mm. The electric stimulators (SDZ-V electroacupuncture apparatus, Suzhou Medical Appliance Factory, China) will connect bilateral BL32, BL33, BL35 and SP 6 and a continuous wave of 10 Hz frequency and an intensity of 0.1-0.3mA will be applied.
  The needles will be retained for 60 mins for each treatment session. The participants will be treated three times a week, on alternate days, for 12 successive weeks; 18 sessions for each patient in total.
  Arms: Sham electroacupuncture

SUMMARY:
Chronic Urinary Retention (CUR) is defined as a non-painful bladder which remains palpable or percussible after the patient has passed urine by International Continence Society. Postvoid residual urine volume ≥300 mL seems to be widely accepted.

CUR may be caused by a variety of diseases and events including injury of sacral plexus, cauda equina and sacral spinal cord, pelvic floor nerve lesion after pelvic surgery and peripheral neuropathy due to diabetes, etc.. Aforementioned injuries generally affect lower motor neuron causing detrusor underactivity, acontractile detrusor or detrusor areflexia. The prevalence varies by different causes of lower motor neuron lesion. The symptoms of patients are voiding difficulty, bladder distention, bladder without sensation and overflow incontinence.

A multi-center randomized sham-controlled trial will be conducted. The aim of this study is to assess the efficacy and safety of electroacupuncture for urinary function of patients with CUR caused by lower motor neuron lesion.

ELIGIBILITY:
Inclusion Criteria:

* Have chronic urinary retention caused by lower motor neuron damage.
* Age 18 to 75 years.
* Have chronic urinary retention caused by injury of sacral plexus, cauda equina and sacral spinal cord, pelvic floor nerve lesion after pelvic surgery and peripheral neuropathy due to diabetes.
* Have postvoid residual urine volume 300 mL or more and sensation of bladder.
* Bladder contractile index is more than 100 or more.
* Duration of disease is more than 3 months.
* Intermittent clean catheterization or indwelling catheterization.
* Sign informed consent and participate in the study voluntarily.
* Exclusion Criteria:
* Have urinary retention due to bladder outlet obstruction (bladder neck contracture, urethral stricture, prostate cancer, prostatic hyperplasia, etc.)
* Have urinary system tumors or stones.
* Have detrusor underactivity due to other non-lower motor neurogenic disease.
* Have bowel and urinary disorder due to lesions or injuries of thoracic spinal cord, cervical spinal cord and brain.
* After suprapubic cystostomy.
* Have heart, liver, kidney, mental disorders or coagulation disorders.
* Have been implanted a cardiac pacemaker, sacral nerve stimulation electrode, pudendal nerve stimulation electrode, or bladder stimulation electrode.
* During pregnancy or in lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-10-09 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The proportions of responders of postvoid residual urine (PVR) | week 12
  The responder is defined as a participant with a decline of 50% or more from baseline in the PVR volume after spontaneous urination. The PVR volume is the average value of 2 times of the same measurement method with the interval of 6 hours to 3 days.

SECONDARY OUTCOMES:
The proportions of responders of postvoid residual urine (PVR) | week 6
  The responder is defined as a participant with a decline of 50% or more from baseline in the PVR volume after spontaneous urination. The PVR volume is the average value of 2 times of the same measurement method with the interval of 6 hours to 3 days.
The proportions of responders of postvoid residual urine (PVR) | week 24
  The responder is defined as a participant with a decline of 50% or more from baseline in the PVR volume after spontaneous urination. The PVR volume is the average value of 2 times of the same measurement method with the interval of 6 hours to 3 days.
The proportions of responders of postvoid residual urine (PVR) | week 36
  The responder is defined as a participant with a decline of 50% or more from baseline in the PVR volume after spontaneous urination. The PVR volume is the average value of 2 times of the same measurement method with the interval of 6 hours to 3 days.
The satisfactory spontaneous urination responders | week 12
  The satisfactory spontaneous urination responders were defined as participants with PVR volume 100 mL or less, without hydronephrosis and recurrent symptomatic urinary tract infection. Recurrent symptomatic urinary tract infection is defined as 2 times or more symptomatic urinary tract infection during the treatment and follow-up period.
The satisfactory spontaneous urination responders | week 24
  The satisfactory spontaneous urination responders were defined as participants with PVR volume 100 mL or less, without hydronephrosis and recurrent symptomatic urinary tract infection. Recurrent symptomatic urinary tract infection is defined as 2 times or more symptomatic urinary tract infection during the treatment and follow-up period.
The satisfactory spontaneous urination responders | week 36
  The satisfactory spontaneous urination responders were defined as participants with PVR volume 100 mL or less, without hydronephrosis and recurrent symptomatic urinary tract infection. Recurrent symptomatic urinary tract infection is defined as 2 times or more symptomatic urinary tract infection during the treatment and follow-up period.
The proportion of patients with increase of 50% or more from baseline of the maximum flow rate (Qmax) | week 12
The proportion of patients with increase of 50% or more from baseline of the maximum flow rate (Qmax) | week 36
The proportion of patients with increase of 2 ml/s from baseline of the maximum flow rate (Qmax) | week 12
The proportion of patients with increase of 2 ml/s from baseline of the maximum flow rate (Qmax) | week 36
The change from baseline of the number of catheterizations per day measured by the 7-day voiding diaries for patients with intermittent clean urethral catheterization | week 6
The change from baseline of the number of catheterizations per day measured by the 7-day voiding diaries for patients with intermittent clean urethral catheterization | week 12
The change from baseline of the number of catheterizations per day measured by the 7-day voiding diaries for patients with intermittent clean urethral catheterization | week 24
The change from baseline of the number of catheterizations per day measured by the 7-day voiding diaries for patients with intermittent clean urethral catheterization | week 36
The proportion of patients with increase of 50% or more from baseline of the voiding efficiency (VE) measured by the 7-day voiding diaries | week 12
  VE is calculated as follows: volume voided/ (volume voided +PVR)*100%
The proportion of patients with increase of 50% or more from baseline of the voiding efficiency (VE) measured by the 7-day voiding diaries | week 36
  VE is calculated as follows: volume voided/ (volume voided +PVR)*100%
The change form baseline of Short Form of a Urinary Quality of Life Questionnaire (SF-Qualiveen) | week 12
  SF-Qualiveen is the only questionnaire that addresses the broad range of urinary problems experienced by patients with neurological disorders voiding symptoms. Qualiveen domain scores are calculated as an average of the scores on items in that domain and, thus, the range is 0 to 4 with an overall score representing the mean of the 4 domains, which also ranges from 0 to 4. A higher score indicates the greater the impact on the quality of life of patients.
The change form baseline of Short Form of a Urinary Quality of Life Questionnaire (SF-Qualiveen) | week 36
  SF-Qualiveen is the only questionnaire that addresses the broad range of urinary problems experienced by patients with neurological disorders voiding symptoms. Qualiveen domain scores are calculated as an average of the scores on items in that domain and, thus, the range is 0 to 4 with an overall score representing the mean of the 4 domains, which also ranges from 0 to 4. A higher score indicates the greater the impact on the quality of life of patients.
The proportion of patients without recurrent symptomatic urinary tract infection, vesical calculus and hydronephrosis | week 12
The proportion of patients without recurrent symptomatic urinary tract infection, vesical calculus and hydronephrosis | week 24
The proportion of patients without recurrent symptomatic urinary tract infection, vesical calculus and hydronephrosis | week 36
The change of the urodynamic parameters from baseline | week 12
  The urodynamic parameters include: bladder capacity (ml), bladder compliance (cmH2O), vesica-open pressure (Pves-open) (cmH2O), maximum flow rate (mL/s), mean flow rate (ml/s), detrusor pressure at maximum flow rate (ml/s), time to maximum flow rate (sec), maximum detrusor pressure (cmH2O), voided volume (ml), residual urine (ml).
The change of the bladder contractile index (BCI) | week 12
  BCI = detrusor pressure at maximum flow rate (Qmax) + 5*Qmax.

OTHER OUTCOMES:
The correlation between expectation assessment and the primary outcome | Baseline
  Expectation assessment will be assessed at baseline; it includes two brief questions to investigate whether patients are confident that acupuncture treatment will help their chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS): "In general, do you believe acupuncture is effective for treating the illness?", "Do you think acupuncture will be helpful to improve your CP/CPPS symptoms?" For each question, participants will choose "Yes", "No", or "unclear" as the answer.
The proportions of participants in each response category of the GRA (Global Response Assessment) in the two groups after treatment | week 12
  GRA consists of 7 response categories: markedly worsened, moderately worsened, slightly worsened, no change, slightly improved, moderately improved, and markedly improved. We will identify a participant who reports "moderate" or "marked improvement" as a responder.
The proportions of participants in each response category of the GRA (Global Response Assessment) in the two groups after treatment | week 24
  GRA consists of 7 response categories: markedly worsened, moderately worsened, slightly worsened, no change, slightly improved, moderately improved, and markedly improved. We will identify a participant who reports "moderate" or "marked improvement" as a responder.
The proportions of participants in each response category of the GRA (Global Response Assessment) in the two groups after treatment | week 36
  GRA consists of 7 response categories: markedly worsened, moderately worsened, slightly worsened, no change, slightly improved, moderately improved, and markedly improved. We will identify a participant who reports "moderate" or "marked improvement" as a responder.
Patient Blinding assessment | week 12
  To test the success of blinding, participants will be asked to reply to the following question at the 12th week of treatment (sessions 35 or 36): "Do you think you have received traditional electroacupuncture in the past weeks?" The participants will be able to choose one of the following options as the answer: "Yes", "No"
Safety assessment | week 1 to week 36
  Treatment-related adverse events (AEs) include pain, haematoma, localized infection, broken needle, fainting, nausea, headache, dizziness, insomnia, vomiting, or palpitations during or after treatment. In addition, adverse events that are irrelevant to the treatment will be recorded during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, PhD, Study Chair — Guang An Men Hospital
Locations (1):
- Guangan'men Hospital, Beijing, China